CLINICAL TRIAL: NCT06462170
Title: The Feasibility of an Innovative Protocol to Demonstrate the Impact of Positive Energy Balance on Pancreatic Insulin Production Capacity (PIPC)
Brief Title: Pancreatic Insulin Production Capacity (PIPC) - a Feasibility Study
Acronym: PIPC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20240236-01H
Record Dates: First submitted 2024-06-07; First posted 2024-06-17 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pancreatic insulin production after drinking meal replacement shake (Experimental): Nutritional intervention, and then blood work will be drawn to measure pancreatic insulin production capacity.
  Interventions: Dietary Supplement: Boost Original meal replacement shake

INTERVENTIONS:
Dietary Supplement: Boost Original meal replacement shake — One bottle of Boost Original meal replacement shake.

SUMMARY:
The standard treatment for Type 2 diabetes involves management of the disease based on average of blood glucose control over the past few months.

In this study, the investigators test for the participants' ability to produce insulin, which is the hormone that the body makes to control blood sugar levels. The body produces insulin in response to eating. The participants will drink a meal replacement shake, and then test the blood for levels of insulin produced over 2 hours.

With blood tests taken five times over two hours, the investigators will measure the blood glucose (sugar), and insulin levels. This study will assess the differences in insulin produced in the participants and try to understand the reasons for these differences.

DETAILED DESCRIPTION:
This study will measure the ability of the pancreas to produce insulin after the participant drinks a Boost Original meal replacement shake. The Boost Original meal replacement shake contains nutrients similar to a typical meal, and allows to standardize this "meal" for all participants. This is a cross-sectional study for 90 participants with type 2 diabetes mellitus who undergo a single study visit that lasts 2 hours with blood drawn at five time points. The area under the curve will be a quantitative measure of each participant's pancreatic insulin production capacity.

ELIGIBILITY:
Inclusion Criteria:

1. Consent provided
2. Age >= 18 years.
3. Diagnosed as type 2 diabetes mellitus.
4. Not on insulin therapy.

Exclusion Criteria:

1. Diagnosed as another form of diabetes mellitus.
2. Allergic to one or more ingredients in Boost meal replacement shake.
3. Unable to fast since midnight and attend in person for the morning protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pancreatic insulin production capacity (PIPC) represented by the participant's insulin and C-peptide levels after drinking the meal replacement shake. | 12 months
  Participants will get blood drawn at time 0, 30, 60, 90, and 120 minutes. Blood will be sent for glucose, insulin, and C-peptide measurements. The area under the curve (AUC) will be calculated from these measurements. The AUC for insulin and for C-peptide will be representative of the participant's PIPC.

SECONDARY OUTCOMES:
The impact of participant's self-reported weight gain in the past year (12 months prior to the single study visit) on participant's PIPC. | 12 months
  Linear regression modelling will be used where weight gain is an independent variable, and PIPC is the dependent variable. The p-value for participant's self-reported weight gain will show the significance of impact on PIPC.

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Sun, MD MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No